CLINICAL TRIAL: NCT05771636
Title: Can Mental Imagery Increase Behavioral Activation ?
Brief Title: Mental Imagery and Psychological Well-being
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Ecaterina Lazari, Principal Investigator, University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1959-827
Record Dates: First submitted 2023-03-01; First posted 2023-03-16 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Depression; Anhedonia
MeSH Terms: conditions — Depression; Anhedonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental G1 - imagery of planned activity (Experimental): In this condition, the participant will have to think about 4 activities he will plan to do during the next 2 weeks. He will then complete a questionnaire about all the activities he identified and think about the major obstacle that could prevent him to do each activity, and a solution for each one. Then he will proceed to a mental imagery exercise where he imagines doing the activity as vividly as possible. He then will proceed to go home and repeat the imagery practice every day for the next two weeks, and do the planned activities. He will report in a booklet ratings of the mental imagery exercise and the activities he did.
  Interventions: Behavioral: Mental Imagery
- Experimental G2 - imagery of best possible self (Experimental): In this condition, the participant will first have to do a mental imagery exercise where he imagines his best possible self, having accomplished all his big life goals, as vividly as possible. He will then have to think about 4 activities he will plan to do during the next 2 weeks, in line with the imagery exercise. He will then complete a questionnaire about all the activities he identified. He then will proceed to go home and repeat the imagery practice every day for the next two weeks, and do the planned activities. He will report in a booklet ratings of the mental imagery exercise and the activities he did.
  Interventions: Behavioral: Mental Imagery
- Control G3 - activity planification alone (Active Comparator): In this condition, the participant will have to think about 4 activities he will plan to do during the next 2 weeks. He will then complete a questionnaire about all the activities he identified. There is no mental imagery exercise in this condition. He then will proceed to go home and receive the assignment to do the planned activities in the course of the next two weeks. He will report in a booklet ratings of the activities he did.
  Interventions: Behavioral: Control condition (activity planification)

INTERVENTIONS:
Behavioral: Mental Imagery — Mental Imagery consists of imagining a situation in the most vivid way possible, including all sensory modalities (visual image, sensations, smells, sounds, emotions). It can be used to act as a motivational amplifier, by pre-experimenting a situation in imagination.
  The best possible self imagery consists of imagining the best version possible of one's self , after accomplishing all their major life goals, in a future where everything turned out the best way possible. What does this best version of you do, in terms of actions, on an everyday basis ? The planned imagery exercise consists of rehearsing an activity in a mental way, before actually doing it. It can help to visualize the outcome of this activity and benefits it can provide to the participant before actually getting it done.
  Arms: Experimental G1 - imagery of planned activity; Experimental G2 - imagery of best possible self
Behavioral: Control condition (activity planification) — The participant identifies 4 activities that he plans to do in the course of the next 2 weeks.
  Arms: Control G3 - activity planification alone

SUMMARY:
This study aims to investigate the effects of mental imagery practice on depression, behavioral activation, psychological well-being and other processes involved in depression such as anhedonia.

We use a multiple baseline design in addition to a pre-post and follow-up standardized assessment design.

DETAILED DESCRIPTION:
The purpose of this study is to determine if daily practice of mental imagery improves psychological variables such as motivation, behavioral activation, depression, mood, optimism, anhedonia, and psychological well-being, and if it's combination with activity planning is more effective than activity planning alone. This study will analyze the effect of 2 mental imagery conditions (planned activity imagery, best possible self) and a control condition of activity planning alone, administered to a general population over a 2-week period.

Our hypotheses are an improvement for both experimental conditions (planned activities imagery and best possible self imagery) of mood, behavioral activation, depressive symptomatology, optimism, psychological well-being, cognitive and behavioral avoidance, and anhedonia, compared to the control condition. Several studies have been able to show the effect of either imagery condition on certain variables (notably behavioral activation and mood for the planned activity imagery as well as optimism and mood for the best possible self), but the interest of our study is to assess the effect of each of the proposed protocols on a broader range of variables. This will allow us to determine the specific effect of each protocol as well as to compare their effectiveness.

In this study we will recruit 120 participants, randomly assigned to one of three conditions: (1) mental imagery of planned activities, (2) mental imagery of best possible self, (3) planned activity control group. All participants will be asked to complete a series of standardized assessments in 4 steps (at the first meeting, at the second meeting 15 days later, and a follow-up at 1 and 3 months post-intervention). The questionnaires will assess depression, behavioral activation, mood, optimism, imagery skills, anhedonia, and psychological well-being.

In each group, participants will have to think about 4 activities to be implemented within the next two weeks, and answer about 10 questions about the chosen activities (rated from 0 to 10 on a visual analogical scale). These questions evaluate, among other things, the motivation, the anticipated effort, the anticipated pleasure, and the degree of avoidance related to each activity using a visual analog scale. This questionnaire will be completed at the first meeting and also after the completion of each activity, at home. The protocol is identical for each condition except for the content of the imagery exercise or no imagery exercise for the control condition. The participants in the experimental conditions will be instructed to repeat the 5-minute imagery exercise at home every day for 2 weeks and report in a booklet everyday their rating of the imagery exercise (vividness, difficulty and their mood after the exercise).

At a second meeting 2 weeks later, all participants will be asked to complete the standardized assessments again and report whether or not the planned activities were completed, as well as conduct a semi-structured interview about their experience, the feasibility and difficulty of the task. Participants will then receive a follow-up survey by e-mail at 1 and 3 months post-intervention, in which they will again be asked to complete the selected standardized questionnaires. The booklets in which they reported the questionnaires about their planned activities (all conditions) and the ratings of imagery exercise (for experimental conditions) will be brought back on that meeting.

ELIGIBILITY:
Inclusion Criteria:

* At least some symptoms of depression (minimal score of 8 on the depression subscale of the HADS)

Exclusion Criteria:

* Not ongoing psychotherapy at the time of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Depressive symptomatology | Baseline
  The Beck depression inventory- second edition (BDI-II) is a 21-items scale that assesses the severity of depressive symptoms during the last two weeks. The score may range from 0 to 63. Higher score indicates higher depressive symptoms (worse outcome).
Depressive symptomatology | Two weeks after beginning of treatment (end of treatment)
  The Beck depression inventory- second edition (BDI-II) is a 21-items scale that assesses the severity of depressive symptoms during the last two weeks. The score may range from 0 to 63. Higher score indicates higher depressive symptoms (worse outcome).
Depressive symptomatology | 1 month after end of treatment
  The Beck depression inventory- second edition (BDI-II) is a 21-items scale that assesses the severity of depressive symptoms during the last two weeks. The score may range from 0 to 63. Higher score indicates higher depressive symptoms (worse outcome).
Depressive symptomatology | 3 months after end of treatment
  The Beck depression inventory- second edition (BDI-II) is a 21-items scale that assesses the severity of depressive symptoms during the last two weeks. The score may range from 0 to 63. Higher score indicates higher depressive symptoms (worse outcome).
Behavioral activation | Baseline
  The Behavioral Activation for Depression Scale (BADS) is a 25-items scale that assesses behavioral activation. Five subscales have been identified: Activation, Behavioral Avoidance, Rumination, Work/School Impairment and Social Impairment. Activation may range from 0 to 42. Higher scores indicate greater activation level (better outcome)
Behavioral activation | Two weeks after beginning of treatment (end of treatment)
  The Behavioral Activation for Depression Scale (BADS) is a 25-items scale that assesses behavioral activation. Five subscales have been identified: Activation, Behavioral Avoidance, Rumination, Work/School Impairment and Social Impairment. Activation may range from 0 to 42. Higher scores indicate greater activation level (better outcome)
Behavioral activation | 1 month after end of treatment
  The Behavioral Activation for Depression Scale (BADS) is a 25-items scale that assesses behavioral activation. Five subscales have been identified: Activation, Behavioral Avoidance, Rumination, Work/School Impairment and Social Impairment. Activation may range from 0 to 42. Higher scores indicate greater activation level (better outcome)
Behavioral activation | 3 months after end of treatment
  The Behavioral Activation for Depression Scale (BADS) is a 25-items scale that assesses behavioral activation. Five subscales have been identified: Activation, Behavioral Avoidance, Rumination, Work/School Impairment and Social Impairment. Activation may range from 0 to 42. Higher scores indicate greater activation level (better outcome)
LOT | Baseline
  The Life Orientation Test (Revised) is a 10-items scale assesses one's dispositional level of optimism, providing meaningful insight into possible interventions, such as those to address harmful thought patterns. Scores can range from 0 to 24, being 0-13 Low Optimism, 14-18 Moderate Optimism, 19-24 High Optimism.
LOT | Two weeks after beginning of treatment (end of treatment)
  The Life Orientation Test (Revised) is a 10-items scale assesses one's dispositional level of optimism, providing meaningful insight into possible interventions, such as those to address harmful thought patterns. Scores can range from 0 to 24, being 0-13 Low Optimism, 14-18 Moderate Optimism, 19-24 High Optimism.
LOT | 1 month after end of treatment
  The Life Orientation Test (Revised) is a 10-items scale assesses one's dispositional level of optimism, providing meaningful insight into possible interventions, such as those to address harmful thought patterns. Scores can range from 0 to 24, being 0-13 Low Optimism, 14-18 Moderate Optimism, 19-24 High Optimism.
LOT | 3 months after end of treatment
  The Life Orientation Test (Revised) is a 10-items scale assesses one's dispositional level of optimism, providing meaningful insight into possible interventions, such as those to address harmful thought patterns. Scores can range from 0 to 24, being 0-13 Low Optimism, 14-18 Moderate Optimism, 19-24 High Optimism.
PANAS | Baseline
  The Positive affect negative affect scale consists of two 10-item scales to measure both positive and negative affect. Each item is rated on a 5-point scale of 1 (not at all) to 5 (very much)
PANAS | Two weeks after beginning of treatment (end of treatment)
  The Positive affect negative affect scale consists of two 10-item scales to measure both positive and negative affect. Each item is rated on a 5-point scale of 1 (not at all) to 5 (very much)
PANAS | 1 month after end of treatment
  The Positive affect negative affect scale consists of two 10-item scales to measure both positive and negative affect. Each item is rated on a 5-point scale of 1 (not at all) to 5 (very much)
PANAS | 3 months after end of treatment
  The Positive affect negative affect scale consists of two 10-item scales to measure both positive and negative affect. Each item is rated on a 5-point scale of 1 (not at all) to 5 (very much).
Anhedonia | Baseline
  The Savoring belief Inventory (SBI) is an 24-items scale assessing individuals' attitudes regarding savoring positive experiences. Three subscales related to three temporal orientations are identified, one related to the past (reminiscence), one related to the present moment (present), and one related to the future (anticipation) each represented by 8 items. Higher scores indicate higher level of approach and savor pleasant events (better outcome).
Anhedonia | Two weeks after beginning of treatment (end of treatment)
  The Savoring belief Inventory (SBI) is an 24-items scale assessing individuals' attitudes regarding savoring positive experiences. Three subscales related to three temporal orientations are identified, one related to the past (reminiscence), one related to the present moment (present), and one related to the future (anticipation) each represented by 8 items. Higher scores indicate higher level of approach and savor pleasant events (better outcome).
Anhedonia | 1 month after end of treatment
  The Savoring belief Inventory (SBI) is an 24-items scale assessing individuals' attitudes regarding savoring positive experiences. Three subscales related to three temporal orientations are identified, one related to the past (reminiscence), one related to the present moment (present), and one related to the future (anticipation) each represented by 8 items. Higher scores indicate higher level of approach and savor pleasant events (better outcome).
Anhedonia | 3 months after end of treatment
  The Savoring belief Inventory (SBI) is an 24-items scale assessing individuals' attitudes regarding savoring positive experiences. Three subscales related to three temporal orientations are identified, one related to the past (reminiscence), one related to the present moment (present), and one related to the future (anticipation) each represented by 8 items. Higher scores indicate higher level of approach and savor pleasant events (better outcome).
Well-being | Baseline
  The Warwick-Edinburgh Mental Well-Being Scale (WEMWBS) is a 14-items scale assessing mental well-being. The score may range from 14 to 70. Higher scores indicate higher mental well-being (better outcome).
Well-being | Two weeks after beginning of treatment (end of treatment)
  The Warwick-Edinburgh Mental Well-Being Scale (WEMWBS) is a 14-items scale assessing mental well-being. The score may range from 14 to 70. Higher scores indicate higher mental well-being (better outcome).
Well-being | 1 month after end of treatment
  The Warwick-Edinburgh Mental Well-Being Scale (WEMWBS) is a 14-items scale assessing mental well-being. The score may range from 14 to 70. Higher scores indicate higher mental well-being (better outcome).
Well-being | 3 months after end of treatment
  The Warwick-Edinburgh Mental Well-Being Scale (WEMWBS) is a 14-items scale assessing mental well-being. The score may range from 14 to 70. Higher scores indicate higher mental well-being (better outcome).
Mental Imagery ability | Baseline
  The Plymouth Sensory Imagery questionnaire is a 35 items scale measuring the vividness of mental imagery in seven different modalities: vision, sound, smell, taste, touch, bodily sensation, and emotion. There is a sub-score for every modality, with score ranging from 5 to 50 (better outcome) and a total score ranging from 35 to 350 (better outcome) higher score indicating higher imagery ability.
Mental Imagery ability | Two weeks after beginning of treatment (end of treatment)
  The Plymouth Sensory Imagery questionnaire is a 35 items scale measuring the vividness of mental imagery in seven different modalities: vision, sound, smell, taste, touch, bodily sensation, and emotion. There is a sub-score for every modality, with score ranging from 5 to 50 (better outcome) and a total score ranging from 35 to 350 (better outcome) higher score indicating higher imagery ability.
Mental Imagery ability | 1 month after end of treatment
  The Plymouth Sensory Imagery questionnaire is a 35 items scale measuring the vividness of mental imagery in seven different modalities: vision, sound, smell, taste, touch, bodily sensation, and emotion. There is a sub-score for every modality, with score ranging from 5 to 50 (better outcome) and a total score ranging from 35 to 350 (better outcome) higher score indicating higher imagery ability.
Mental Imagery ability | 3 months after end of treatment
  The Plymouth Sensory Imagery questionnaire is a 35 items scale measuring the vividness of mental imagery in seven different modalities: vision, sound, smell, taste, touch, bodily sensation, and emotion. There is a sub-score for every modality, with score ranging from 5 to 50 (better outcome) and a total score ranging from 35 to 350 (better outcome) higher score indicating higher imagery ability.

SECONDARY OUTCOMES:
self concordant motivation | Baseline
  The self concordance motivation scale is a scale in which the participant rates his motivation to pursue a goal based on 4 different reasons (external, introjected, identified and intrinsic) on a scale from 1 to 9, designed to measure if the motivation of a person relative to his goals is intrinsic or extrinsic.
  The self-concordance variable is calculated by averaging the intrinsic and identified ratings and subtracting the average external and introjected ratings. A higher score means higher self-concordance (better outcome)
Motivation to do this activity | Baseline
  Assessment on a scale from 0 (minimum, worse outcome) to 10 (maximum, better outcome) of the effects and costs of this activity perceived by the participant. The question is asked for each identified activity.
Motivation to do this activity | Right before doing the activity (during the two weeks intervention, reporting in the booklet, at home)
  Assessment on a scale from 0 (minimum, worse outcome) to 10 (maximum, better outcome) of the effects and costs of this activity perceived by the participant. The question is asked for each identified activity.
Positive anticipation of the activity | Baseline
  Assessment on a scale from 0 (minimum, worse outcome) to 10 (maximum, better outcome) of the effects and costs of this activity perceived by the participant. The question is asked for each identified activity.
Positive anticipation of the activity | Right before doing the activity (during the two weeks intervention, reporting in the booklet, at home)
  Assessment on a scale from 0 (minimum, worse outcome) to 10 (maximum, better outcome) of the effects and costs of this activity perceived by the participant. The question is asked for each identified activity.
Anticipated pleasure resulting in the activity | Baseline
  Assessment on a scale from 0 (minimum, worse outcome) to 10 (maximum, better outcome) of the effects and costs of this activity perceived by the participant. The question is asked for each identified activity.
Anticipated pleasure resulting in the activity | Right before doing the activity (during the two weeks intervention, reporting in the booklet, at home)
  Assessment on a scale from 0 (minimum, worse outcome) to 10 (maximum, better outcome) of the effects and costs of this activity perceived by the participant. The question is asked for each identified activity.
Anticipated satisfaction resulting in the activity | Baseline
  Assessment on a scale from 0 (minimum, worse outcome) to 10 (maximum, better outcome) of the effects and costs of this activity perceived by the participant. The question is asked for each identified activity.
Anticipated satisfaction resulting in the activity | Right before doing the activity (during the two weeks intervention, reporting in the booklet, at home)
  Assessment on a scale from 0 (minimum, worse outcome) to 10 (maximum, better outcome) of the effects and costs of this activity perceived by the participant. The question is asked for each identified activity.
Anticipated Gratification resulting in the activity | Baseline
  Assessment on a scale from 0 (minimum, worse outcome) to 10 (maximum, better outcome) of the effects and costs of this activity perceived by the participant. The question is asked for each identified activity.
Anticipated Gratification resulting in the activity | Right before doing the activity (during the two weeks intervention, reporting in the booklet, at home)
  Assessment on a scale from 0 (minimum, worse outcome) to 10 (maximum, better outcome) of the effects and costs of this activity perceived by the participant. The question is asked for each identified activity.
Anticipated difficulty to do the activity | Baseline
  Assessment on a scale from 0 (minimum, better outcome) to 10 (maximum, worse outcome) of the effects and costs of this activity perceived by the participant. The question is asked for each identified activity.
Anticipated difficulty to do the activity | Right before doing the activity (during the two weeks intervention, reporting in the booklet, at home)
  Assessment on a scale from 0 (minimum, better outcome) to 10 (maximum, worse outcome) of the effects and costs of this activity perceived by the participant. The question is asked for each identified activity.
Avoidance of the activity | Baseline
  Assessment on a scale from 0 (minimum, better outcome) to 10 (maximum, worse outcome) of the effects and costs of this activity perceived by the participant. The question is asked for each identified activity.
Avoidance of the activity | Right before doing the activity (during the two weeks intervention, reporting in the booklet, at home)
  Assessment on a scale from 0 (minimum, better outcome) to 10 (maximum, worse outcome) of the effects and costs of this activity perceived by the participant. The question is asked for each identified activity.
Importance of the activity | Baseline
  Assessment on a scale from 0 (minimum, worse outcome) to 10 (maximum, better outcome) of the effects and costs of this activity perceived by the participant. The question is asked for each identified activity.
Importance of the activity | Right before doing the activity (during the two weeks intervention, reporting in the booklet, at home)
  Assessment on a scale from 0 (minimum, worse outcome) to 10 (maximum, better outcome) of the effects and costs of this activity perceived by the participant. The question is asked for each identified activity.
Difficulty to find time to do the activity | Baseline
  Assessment on a scale from 0 (minimum, better outcome) to 10 (maximum, worse outcome) of the effects and costs of this activity perceived by the participant. The question is asked for each identified activity.
Difficulty to find time to do the activity | Right before doing the activity (during the two weeks intervention, reporting in the booklet, at home)
  Assessment on a scale from 0 (minimum, better outcome) to 10 (maximum, worse outcome) of the effects and costs of this activity perceived by the participant. The question is asked for each identified activity.
Perceived difficulty after doing the activity | Right after doing the activity (during the two weeks intervention, reporting in the booklet, at home)
  Assessment on a scale from 0 (minimum, worse outcome) to 10 (maximum, better outcome) of the effects and costs of this activity perceived by the participant. The question is asked for each identified activity.
Perceived mood after doing the activity | Right after doing the activity (during the two weeks intervention, reporting in the booklet, at home)
  Assessment on a scale from 0 (minimum, worse outcome) to 10 (maximum, better outcome) of the effects and costs of this activity perceived by the participant. The question is asked for each identified activity.
Perceived pleasure after doing the activity | Right after doing the activity (during the two weeks intervention, reporting in the booklet, at home)
  Assessment on a scale from 0 (minimum, worse outcome) to 10 (maximum, better outcome) of the effects and costs of this activity perceived by the participant. The question is asked for each identified activity.
Perceived satisfaction after doing the activity | Right after doing the activity (during the two weeks intervention, reporting in the booklet, at home)
  Assessment on a scale from 0 (minimum, worse outcome) to 10 (maximum, better outcome) of the effects and costs of this activity perceived by the participant. The question is asked for each identified activity.
Perceived gratification after doing the activity | Right after doing the activity (during the two weeks intervention, reporting in the booklet, at home)
  Assessment on a scale from 0 (minimum, worse outcome) to 10 (maximum, better outcome) of the effects and costs of this activity perceived by the participant. The question is asked for each identified activity.
Difficulty of the mental imagery exercise | Everyday at home during the two weeks intervention period, right after doing the imagery exercise (reporting in the booklet, at home)
  Assessment on a scale from 0 (minimum, worse outcome) to 10 (maximum, better outcome) of the effects and costs of this activity perceived by the participant. The question is asked for each identified activity.
Mood after doing the mental imagery exercise | Everyday at home during the two weeks intervention period, right after doing the imagery exercise (reporting in the booklet, at home)
  Assessment on a scale from 0 (minimum, worse outcome) to 10 (maximum, better outcome) of the effects and costs of this activity perceived by the participant. The question is asked for each identified activity.
Vividness of the mental imagery exercise | Everyday at home during the two weeks intervention period, right after doing the imagery exercise (reporting in the booklet, at home)
  Assessment on a scale from 0 (minimum, worse outcome) to 10 (maximum, better outcome) of the effects and costs of this activity perceived by the participant. The question is asked for each identified activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Université de Liège, Liège, Belgium